CLINICAL TRIAL: NCT06118476
Title: The Effect of Education Provided to Nursing Students With 3D Animation on Course
Brief Title: The Effect of Education Provided to Nursing Students With 3D Animation on Course Interest, Motivation and Attitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Metin Yildiz, Nurse (Asst.Prof.Dr.), Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SakaryaU-metinyildiz-006
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Educational Problems
Keywords: 3D Animation; Interest; Motivation; Attitude to the Course

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group trained with 3D animation (Experimental): The experimental group was followed by training with 3D animation videos every week.
  Interventions: Behavioral: 3D animation
- Control group (No Intervention): Lessons were taught with traditional learning method.

INTERVENTIONS:
Behavioral: 3D animation — Education with 3D animation videos
  Arms: Group trained with 3D animation

SUMMARY:
Along with traditional education methods, it is important to try different methods in order to increase interest, attitude and motivation in the lesson in accordance with the requirements of the age. Our study aimed to examine nursing students' attitudes towards the course in line with the principle of attractiveness in education. The study was conducted between March 2023 and June. The population of the research consists of second year students of Sakarya University, Faculty of Health Sciences, Department of Nursing. In the study, randomization determined which of the branches would be the experimental and control group. The sample of the study consisted of all volunteer students. The experimental group was completed with n:60 and the control group with n:57 students. To ensure homogeneity in the study, care was taken to include different branches in the same class. For consistency between observers, it was conducted in a course conducted by the same instructor. Data collection was conducted online. Participants answered the questions of the introductory information form, Instructional Material Motivation Scale, Course Interest Scale, and Attitude Towards Learning Scale. The post-test was administered to the control group without any intervention. The experimental group was trained and monitored with 3D animation videos every week. The data were evaluated using the IBM SPSS Statistics 23 program.

DETAILED DESCRIPTION:
Path Followed in the Study:

Week 1: Separation of Branches randomly Week 1: Experimental and Control Group Pretest Week 6: Final Test after the last training

Data collection tools used in the study:

1. Introductory information form: It consists of questions regarding the demographic characteristics of the students.
2. Instructional Material Motivation Scale (IMMS) The Instructional Material Motivation Scale (IMMS), developed by Keller (2010) and adapted into Turkish by Dinçer et al. (2016), was developed to measure the effect of teaching materials on students' motivation. The original language of the scale is English. In Keller's original IMMS scale, some of the items were designed as positive and some as negative. Accordingly, items 3, 7, 12, 15, 19, 22, 26, 29, 31 and 34 of the scale (10 items in total) are negative; Other items are positive. IMMS scale is a Likert-type scale consisting of 36 items. Each item on the scale will be scored by students from 1 (Not True) to 5 (Very True). Accordingly, the lowest score on the scale is 36 and the highest score is 180. In the reliability analysis, the reliability coefficient (Cronbach Alpha value) was found to be 0.92.
3. Course Interest Scale: Student interest; Course Interest Scale, which was developed to evaluate its relationship with variables such as learning motivation, effective learning, and class participation level, is a 5-point Likert-type measurement tool consisting of 16 items and two sub-dimensions (affective and cognitive interest). The study was adapted by Akın et al. (2015) ( "1" I totally disagree, "2" I disagree, "3" I am undecided, "4" I agree, "5" I totally agree). There are no reverse coded items in the scale. The highest and lowest scores that can be obtained from the scale are 45 and 9, respectively, for the affective interest sub-dimension; 35 and 7 for the cognitive interest sub-dimension. As a result of the analyses, a two-dimensional structure was obtained with factor loadings ranging between .73 and .90. The affective interest sub-dimension of the scale consists of 9 items and the cognitive interest sub-dimension consists of 7 items. Cronbach's alpha internal consistency reliability coefficients of the scale were found to be .95 for the affective interest sub-dimension and .88 for the cognitive interest sub-dimension.
4. Attitude Scale towards Learning (ASTL): The scale developed by Çetin et al. was developed to determine the attitudes of students. As a result of all validity and reliability analyses, ASTL includes a total of 34 items. Of these scale items, 25 are positive and 9 are negative. The scale, which is graded in a five-point Likert style, is "Totally Agree", "To a Great extent", "Partly Agree", "I Disagree", "Totally Disagree". The highest attitude score that can be obtained from the scale is 170 and the lowest attitude score is 34. The 9 negative items in the scale are reverse scored. The Cronbach Alpha internal consistency coefficient of the scale was found to be 0.94 for the overall scale.

In the analysis of data; percentile distribution, chi-square, Fisher- Exact test, t-test in independent groups, paired samples t Test were used.

ELIGIBILITY:
Inclusion Criteria:

2nd year nursing student 18 years and over Voluntarily

Exclusion Criteria:

Students who are not required to attend the course are not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Teaching Material Motivation Scale | Evaluated at the end of 6 weeks
  Teaching Material Motivation Scale Teaching Material Motivation Instructional Material Motivation Scale: It was developed to measure the effect of instructional materials on students' motivation. The scale is a 5-point Likert-type scale consisting of 36 items. Each item in the scale will be scored from 1 (Not True) to 5 (Very True) by the students. Accordingly, the lowest score on the scale is 36, and the highest score is 180. An increase in the score on the scale indicates an increase in motivation.
Course interest scale | Evaluated at the end of 6 weeks
  Developed by (Mazer, 2013) in order to evaluate its relationship with variables such as learning motivation, effective learning, and level of participation in the lesson, the Class Interest Scale is a 5-point Likert-type measurement tool consisting of 16 items and two sub-dimensions (affective and cognitive interest). et al (2015) ("1" Strongly disagree, "2" Disagree, "3" Undecided, "4" Agree, "5" Totally Agree). There is no reverse coded item in the scale. Affective interest sub-dimension of the scale consists of 9 items and cognitive interest sub-dimension consists of 7 items. As the scale score increases, the interest increases.
Attitude Scale Towards Learning | Evaluated at the end of 6 weeks
  Attitude Scale Towards Learning:Attitude Scale Towards Learning: The scale developed by Çetin et al. was developed to determine students' attitudes. As a result of all validity and reliability analyzes, there are 34 items in total. Of these scale items, 25 are positive and 9 are negative. The five-point Likert scale is "Totally Agree", "Strongly Agree", "Partly Agree", "Disagree", "Strongly Disagree". The highest attitude score that can be obtained from the scale is 170 and the lowest attitude score is 34. As the attitude score increases, the positive attitude increases

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)